CLINICAL TRIAL: NCT04355078
Title: Effectiveness of Neuromuscular Training on Lower Extremity in Post-operative Anterior Cruciate Ligament Reconstruction
Brief Title: Neuromuscular Training on Lower Extremity in Post-operative Anterior Cruciate Ligament Reconstruction
Acronym: ENTACLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00587 Kehkshan Khalid
Record Dates: First submitted 2020-02-28; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Anterior cruciate ligament, Neuromuscular training,Strength
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training (Experimental): The rehabilitation program starts two months after surgery, 45 minutes daily session, 3 times a week for 6 weeks. The involved leg is used if nothing else is stated that includes Walking on a treadmill, Squatting exercises, Single leg stance exercise Balance reach leg and arm exercises, Lunge exercises: anterior, lateral and posterior, Step-up and step down exercises, Single leg standing on balance mat, appropriate knee and hip position, Backwards and sideways walking for 5 steps on each side 1, 1 leg and 2 leg Wobble board Exercise and progress after every two weeks
  Interventions: Other: Neuromuscular Training
- Strength Training (Experimental): The rehabilitation program starts two months after surgery, 45 minutes daily session, 3 times a week for 6 weeks that includes straight leg raising exercises, Supine position-isometric quadriceps contraction, Supine position-knee flexion and extension ROM exercises, the heel in contact with the bench during the ROM, Prone position-straight leg raising exercises, Prone position-knee flexion & Extension ROM exercises, Stationary biking-before reaching 100 degrees of flexion(Progression: stair climbing and strength exercises), Standing-full weight-bearing, controlled balance double-limb support during parallel and diagonal stance, controlled knee extension, emphasis on full knee extension in weight-bearing position 3 10 reps Standing heel rising exercises both legs and one leg, 1 leg and 2 leg Wobble board Exercise, Step Up and down low height, Squatting exercises without bars/weight, Hamstrings, hip adductor and abductor strengthening exercises and progress after every two weeks
  Interventions: Other: Strength Training

INTERVENTIONS:
Other: Neuromuscular Training — Muscular and neural training by complex exercises
  Arms: Neuromuscular Training
Other: Strength Training — Strength Training
  Arms: Strength Training

SUMMARY:
The objective of the study was to determine the effectiveness of neuromuscular physical Therapy as compared to strength training after ACL reconstruction in terms of pain, function, quality of life, strength and power of participants after ACL reconstruction.

It was a Randomized clinical trial conducted Kanaan Physiotherapy & Spine Clinic, Lahore. Seventy-six patients were selected by purposive sampling technique and equally divided into one of two treatment groups either neuromuscular training or strength training with use of sealed envelope randomization. The study was completed in 6 months. Patients were assessed using the Cincinnati Knee Score for function, Numeric Pain Rating Scale (NPRS) for pain, SF-36 for quality of life, and Hop test (single leg, Triple, crossover and 6-meter hop) for power and strength.Patients received the treatment 3 times per week for six consecutive weeks.

DETAILED DESCRIPTION:
The knee joint problems and injuries has been rising as a result of more number of patients getting injuries in various daily livings e.g traffic and industrial accidents Ligamentous injuries are one of the commonest injuries of knee among which occurrence of Anterior cruciate ligament(ACL) injuries are of considerable importance The ACL is actually made up of many bundles of connective tissue and it has course from femur to tibia as shown in picture. The ACL is main ligament which prevents tibia to go outwards and excessive loads. When knee is in straight position ACL has 32mm length and 7-12mm width.ACL has 2 parts anteromedial bundle and posterolateral bundle. During flex position AMB goes into lengthened position and PLB goes into shorten position. It is made up of collagen fibres and its framework has proteins, glycoproteins, elastic systems, and glycoseminoglycans. Because of its elastic property it undergoes into many stresses. And it has nerve supply of tibial nerve and it has arterial supply of middle genicular artery. The Occurrence of ACL injures mostly reported among paediatric and adolescent population as compared to adult population. This factor which raises the contribution of adults to participate in sports are younger age high performance training, awareness of injury and use of better modalities. Short term complications of ACL that include loss of function, pain and reconstructive surgery period of about 24 to 36 weeks required for return to function. Reconstructive surgeries include autogenous or allogeneic graft reconstruction Many studies showed that after reconstructive surgery patients return to sports. Most (82%) patients are able to return to sport activity according to a meta-analysis results; however preinjury levels of performance are attained in only 43-65.7% of cases. Long-term complication of ACL injuries that significantly include osteoarthritis that develop later in life. One of the studies show that 50% of diagnosed patients of meniscus or ACL tear might develop osteoarthritis (OA) in the affected knee in about 10-20 years after surgery and the prevalence and severity of OA has not been shown to reduce by reconstructive surgery. Newer surgical approaches and techniques seems to reduce risk of developing osteoarthritis later in life but still questionable.

ELIGIBILITY:
Inclusion Criteria:

* Patients between ages 20-40 years having unilateral ACL injury.
* Patients of both genders.
* Underwent surgical reconstruction of the ACL.
* Participants after two months of ACL unilateral reconstruction.
* Participants who attended physical therapy sessions for first two months to reduce swelling and to gain ROM post operatively.
* Patients willing to participate in the study

Exclusion Criteria:

* History of previous complicated knee surgery
* Non-operative treatment; partial ACL tear; bilateral ACL injury; associated ligament pathology that required surgical treatment at the time of the index surgery; Outerbridge grade III or IV chondral injury; revision ACL reconstruction
* Participation in other studies that may conflict with participation in this study.
* Complex associated injuries (multiple ligamentous injury, extensive cartilage/meniscus injury)
* Recently re-injured in 1 month. Complications such as cancer, inflammatory arthritis, disorders of autoimmune nature (Rheumatoid arthritis), anticoagulant conditions, neurodegenerative diseases (Parkinson's Disease, Motor neuron disease), organic referred pain, pregnancy, and disability compensation.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
NPRS | 4 months
  To rate pain of patients and 1 to 3 considered as mild, 4 to 7 considered as Moderate and 8 to 10 considered as severe pain
SF-36 | 4 months
  Quality of Life

SECONDARY OUTCOMES:
Cincinnati Knee score | 4 months
  The Cincinnati Knee Rating System is one of the most commonly used instruments to measure the results of anterior cruciate ligament reconstruction,The total score is calculated as the sum of all questions responses, with 100 representing the best/excellent knee function, and 0 representing the worst/poor knee function.
Hop Tests | 4 months
  A series of hop tests are routinely used in the assessment for return to sports post-injury, be it an ankle sprain, stress fracture or anterior cruciate ligament reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faheem Afzal, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shim JK, Choi HS, Shin JH. Effects of neuromuscular training on knee joint stability after anterior cruciate ligament reconstruction. J Phys Ther Sci. 2015 Dec;27(12):3613-7. doi: 10.1589/jpts.27.3613. Epub 2015 Dec 28. PMID 26834316
- [Background] Ucar M, Koca I, Eroglu M, Eroglu S, Sarp U, Arik HO, Yetisgin A. Evaluation of open and closed kinetic chain exercises in rehabilitation following anterior cruciate ligament reconstruction. J Phys Ther Sci. 2014 Dec;26(12):1875-8. doi: 10.1589/jpts.26.1875. Epub 2014 Dec 25. PMID 25540486
- [Background] Mather RC 3rd, Hettrich CM, Dunn WR, Cole BJ, Bach BR Jr, Huston LJ, Reinke EK, Spindler KP. Cost-Effectiveness Analysis of Early Reconstruction Versus Rehabilitation and Delayed Reconstruction for Anterior Cruciate Ligament Tears. Am J Sports Med. 2014 Jul;42(7):1583-91. doi: 10.1177/0363546514530866. Epub 2014 May 6. PMID 24801663
- [Background] Risberg MA, Holm I, Myklebust G, Engebretsen L. Neuromuscular training versus strength training during first 6 months after anterior cruciate ligament reconstruction: a randomized clinical trial. Phys Ther. 2007 Jun;87(6):737-50. doi: 10.2522/ptj.20060041. Epub 2007 Apr 18. PMID 17442840
- [Background] Porter MD, Shadbolt B. "Anatomic" single-bundle anterior cruciate ligament reconstruction reduces both anterior translation and internal rotation during the pivot shift. Am J Sports Med. 2014 Dec;42(12):2948-54. doi: 10.1177/0363546514549938. Epub 2014 Sep 19. PMID 25239931
- [Background] Murray JJ, Renier CM, Ahern JJ, Elliott BA. Neuromuscular Training Availability and Efficacy in Preventing Anterior Cruciate Ligament Injury in High School Sports: A Retrospective Cohort Study. Clin J Sport Med. 2017 Nov;27(6):524-529. doi: 10.1097/JSM.0000000000000398. PMID 27755010
- [Background] Struewer J, Frangen TM, Ishaque B, Bliemel C, Efe T, Ruchholtz S, Ziring E. Knee function and prevalence of osteoarthritis after isolated anterior cruciate ligament reconstruction using bone-patellar tendon-bone graft: long-term follow-up. Int Orthop. 2012 Jan;36(1):171-7. doi: 10.1007/s00264-011-1345-0. Epub 2011 Sep 7. PMID 21898038